CLINICAL TRIAL: NCT00316186
Title: An Open-label Phase II Study of Weekly Intravenous Hycamtin and Carboplatin as First-line Treatment of Chemonaive Subjects With Extensive Disease Small Cell Lung Cancer
Brief Title: First-line Treatment Of Subjects With Extensive Disease Small Cell Lung Cancer With Weekly Hycamtin And Paraplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104864/903
Record Dates: First submitted 2006-04-19; First posted 2006-04-20 (Estimated); Results first posted 2009-09-29 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Lung Cancer, Small Cell
Keywords: chemonaive; small cell lung cancer; untreated; Lung cancer; HYCAMTIN; first-line; extensive disease
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Topotecan; Carboplatin

ARMS (1):
- Single arm, open label (Experimental)
  Interventions: Drug: topotecan; Drug: carboplatin

INTERVENTIONS:
Drug: topotecan — Hycamtin and Carboplatin as first-line treatment of chemonaive subjects with EX-SCLC.
Drug: carboplatin — Hycamtin and Carboplatin as first-line treatment of chemonaive subjects with EX-SCLC.
  Other Names: topotecan

SUMMARY:
This study was designed to find the safest and most effective dose of a combination of two chemotherapy drugs, Hycamtin® (topotecan) and Paraplatin® (carboplatin), in people with extensive disease small cell lung cancer.

ELIGIBILITY:
Inclusion criteria:

* Adequate contraception methods include: systemic contraceptives or IUD for 3 months prior to start of the study medication or diaphragm plus spermicide; for males, condom plus spermicide; or total abstinence from sexual intercourse during the course of the study
* Women of childbearing potential and sexually active males must practice or use an accepted and effective form of contraception
* Subjects who present with CNS metastases are eligible, provided the attending physician ascertains that the metastases are controlled before the start of chemotherapy, and the subject is asymptomatic on neurologic exam and is not receiving corticosteroid therapy to control symptoms. Continued use of other anti-seizure medication is permitted
* Free of active infection
* At screening, a probable life expectancy of at least 3 months
* No prior chemotherapy for SCLC or any chemotherapy within 5 years of the diagnosis of SCLC. Prior radiation to any symptomatic site is permitted provided that the indicator lesion site(s) are not irradiated, and radiation is completed before chemotherapy is started
* Performance status ECOG 0-1
* Adequate hematologic, renal and hepatic function •Hematologic: ANC 1500/mm3 [1.5 x 109/L], platelet count 100,000/L (100 x 109/L), hemoglobin 9.0 g/dL
* Renal: Serum Creatinine ≤1.5mg/dL (133mol/L) and CrCl 60 ml/min (Cockroft-Gault) [Cockroft, 1976]

CrCl may be calculated using the Cockcroft-Gault formula:

CrCl (ml/min) = Q x (140-age [yr]) x body wt [kg] 72 x serum creatinine [mg/dl] Q = 0.85 for females Q = 1.0 for males CrCl (ml/min) = K x (140-age [yr]) x body wt [kg] Serum creatinine [mol/L] K = 1.0 for females K = 1.23 for males

* Hepatic: Serum bilirubin (1.5 mg/dL), SGOT (AST), SGPT (ALT) and Alkaline Phosphatase 2 times the upper limit of normal (ULN) if liver metastases are absent by abdominal CT or MRI, or 5 times ULN if liver metastases are present
* At least 18 years old
* Written informed consent (subject's written understanding of and agreement to participate in this study.
* Subject with histologically-confirmed extensive small cell lung cancer or unequivocally positive positive cytological evidence (sputum, at least two, or aspirate biopsy)
* Presence of measurable disease according to World Health Organization (WHO)* criteria, as determined by diagnostic tests, including CT scan of the chest and abdomen, or MRI scan of the brain, or CXR, or PET CT, MRI, and/or CXR are the preferred diagnostic methods to evaluate disease during the course of this study. Use of positron-emission tomography (PET) is not required, but is permitted if it is the standard diagnostic tool employed by the institution. Measurable disease - Presence of at least one bidimensionally measurable, non-CNS lesion (indicator lesion). If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology • Measurable disease, either on CT or MRI scan, requires one diameter 1 cm and one diameter 2 cm. • Measurable disease on CXR requires both diameters 2 cm. • Palpable tumor masses that could not be evaluated radiologically require two diameters 2 cm
* At least 3 weeks since last major surgery (a lesser period is acceptable if decided to be in the best interest of the subject).
* Subjects with central nervous system metastases are eligible as long as the attending doctor determines that the metastases are under control before the start of chemotherapy, and the subject has no symptoms of spreading of disease to the brain, and is not receiving drugs called steroids to control the symptoms.
* Laboratory criteria: Subjects must have adequate bone marrow reserve and adequate kidney and liver function.

Exclusion criteria:

* Concurrent or planned chemotherapy, immunotherapy, radiotherapy, or investigational therapy for the treatment of SCLC. (Concurrent radiation for palliation of bone metastases and CNS lesions must be discussed with and approved by the GlaxoSmithKline Medical Monitor)
* Concurrent severe medical problems other than the diagnosis of SCLC, which would significantly limit full compliance with the study or expose the patient to extreme risk
* Concomitant malignancies or previous malignancies other than SCLC within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or localized low grade prostate cancer (contact GlaxoSmithKline Medical Monitor to discuss enrolment of subjects with low grade prostate cancer)
* Present clinical signs or symptoms of brain and/or leptomeningeal metastases confirmed by CT or MRI brain scan, or corticosteroid treatment to control symptoms of brain metastases
* Uncontrolled infection
* Ongoing tumor or previous tumor other than lung cancer within the last 5 years.
* Symptoms of spreading of the disease to the brain that requires treatment with drugs called steroids
* Severe medical problems other than the diagnosis of SCLC that would limit the ability of the subject to follow study plan or that would expose the subject to extreme risk.
* Ongoing or planned chemotherapy, immunotherapy, radiation treatment, or other experimental drug therapy for the treatment of SCLC.
* Use of investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
* Women who are pregnant or lactating.
* Women who can become pregnant who refuse to practice an adequate form of birth control.
* Subjects with history of allergic reaction to chemicals related to HYCAMTIN and PARAPLATIN.
* Subjects with pre-existing heart disease, such as congestive heart failure, irregular heartbeats that require treatment, and heart attack within the last 3-months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (12):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Munster, Indiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Richmond, Virginia
- GSK Investigational Site, Poznan, Poland

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Topotecan and Carboplatin: Administered Weekly (Days 1 and 8 for topotecan; Day 1 for carboplatin) every 21 days
Period: Overall Study
Arm/Group | Intravenous Topotecan and Carboplatin
Started | 33
Completed | 21
Not Completed | 12
Not completed — Adverse Event | 6
Not completed — Disease Progression | 4
Not completed — Lost to Follow-up | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, as Determined by Radiologic Evaluation (Utilizing the World Health Organization [WHO] Criteria), Calculated as the Number of Participants With the Indicated Response
Description: The categories of tumor response were: complete response (complete disappearance of all known lesions determined by 2 measurements not less than 4 weeks apart), partial response (>50% decrease in measurable lesions for at least 4 weeks with no appearance of new lesions), stable disease (no change in tumor size for at least 8 weeks), progressive disease (>25% increase in measurements of lesions or appearance of new lesions), and not evaluable. The overall response rate was determined using a scan performed within the first 30 days of the first response.
Time Frame: Baseline until up to Day 169
Population: ITT (Intent to Treat): participants that received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 33
Participants
  Complete Response | 0
  Partial Response | 8
  Stable Disease | 11
  Progressive Disease | 6
  Not Evaluable | 8

2. Secondary Outcome: Time to Response
Description: Time to response is calculated as the time from the start of treatment until first documented evidence of partial or complete response. The study was terminated after the dose-finding run-in component was completed because of slow recruitment and acknowledgement of a competing Phase II study. Data not available, as the activity stage was not done.
Time Frame: From start of treatment to evidence of partial or complete response
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Duration
Description: Duration of response is calculated as the time from first documented partial or complete response until first documented sign of disease progression or death. The study was terminated after the dose-finding run-in component was completed because of slow recruitment and acknowledgement of a competing Phase II study. Data not available.
Time Frame: From time of partial or complete response to disease progression/death
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression
Description: Time to progression is defined as the time from the start of treatment until the first documented sign of disease progression or death due to any cause, if sooner. The study was terminated after the dose-finding run-in component was completed because of slow recruitment and acknowledgement of a competing Phase II study. Data not available.
Time Frame: From start of treatment to disease progression/death
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival, Calculated as the Number of Subjects Who Died From the Start of Treatment Until Follow-up
Description: Overall survival is defined as the time from the start of treatment until death due to any cause. The study was terminated after the dose-finding run-in component was completed because of slow recruitment and acknowledgement of a competing Phase II study. Data not available, as the activity stage of the study was not conducted.
Time Frame: Week 1 up to maximum of Day 519
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 0

6. Secondary Outcome: Grade 1 (Mild) Hematological Toxicities
Description: Hematology evaluation included hemoglobin, hematocrit, red blood cell count, white blood cell with differential and platelet count. Differential included neutrophils, bands, lymphocytes, monocytes, eosinophils, and basophils. The intensity of each hematological toxicity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAEs). Hematological toxicities are summarized by Common Terminology Criteria (CTC) V3.0 Maximum Toxicity Grade.
Time Frame: Week 1 through Endpoint (variable based on disease progression or toxicity)
Population: ITT Population (i.e., participants who had at least one dose of study medication)
Measure: Number; unit: participants
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 32
participants
  Anemia | 12
  Neutropenia | 1
  Thrombocytopenia | 15
  Leukopenia | 13

7. Secondary Outcome: Grade 2 (Moderate) Hematological Toxicities
Description: as for outcome 6
Time Frame: Week 1 through Endpoint (variable based on disease progression or toxicity
Population: ITT Population (i.e., participants who had at least one dose of study medication)
Measure: Number; unit: participants
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 32
participants
  Anemia | 14
  Neutropenia | 4
  Thrombocytopenia | 5
  Leukopenia | 10

8. Secondary Outcome: Grade 3 (Severe) Hematological Toxicities
Description: as for outcome 6
Time Frame: Week 1 through Endpoint (variable based on disease progression or toxicity
Population: ITT population (i.e., participants who had at least one dose of study medication)
Measure: Number; unit: participants
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 32
participants
  Anemia | 4
  Neutropenia | 4
  Thrombocytopenia | 2
  Leukopenia | 4

9. Secondary Outcome: Grade 4 (Life-threatening or Disabling) Hematological Toxicities
Description: as for outcome 6
Time Frame: Week 1 through Endpoint (variable based on disease progression or toxicity
Population: ITT population (i.e., participants who had at least one dose of study medication)
Measure: Number; unit: participants
Arm/Group | Intravenous Topotecan and Carboplatin
Number analyzed (Participants) | 32
participants
  Anemia | 2
  Neutropenia | 4
  Thrombocytopenia | 2
  Leukopenia | 0

ADVERSE EVENTS:
Arm/Group | Intravenous Topotecan and Carboplatin
Serious Adverse Events (participants affected / at risk) | 6/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Topotecan and Carboplatin (N=33)
Gastro-intestinal hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Brain Mass (Nervous system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Diease under study (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Topotecan and Carboplatin (N=33)
Anemia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 4
Mucosal inflammation (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 3
Pyrexia (General disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Cardiac disorders) | 2
Dyspnea exertional (Cardiac disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Back Pain (General disorders) | 2
Insomnia (Psychiatric disorders) | 2
Vision Blurred (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.